CLINICAL TRIAL: NCT03091153
Title: Impact of a Deprescribing Intervention on Nursing Home Residents: a Randomized Controlled Trial
Brief Title: Deprescribing in a Long Term Care Facility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Collaborators: Eastern Health (Other)
Responsible Party: Principal Investigator, Deborah Kelly, Associate Professor, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HREB - 2016.312
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Polypharmacy
MeSH Terms: interventions — Medication Review

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard care. Annual medication review
- Intervention (Experimental): In depth medication review with a focus on deprescribing
  Interventions: Other: Medication Review

INTERVENTIONS:
Other: Medication Review — In depth medication review with a focus on deprescribing
  Arms: Intervention

SUMMARY:
This study will develop, implement and evaluate a deprescribing initiative at a Canadian Long Term Care (LTC) Facility. Residents currently undergo an annual medication review as part of the clinical pharmacy services provided in the LTC facility. For this study, eligible residents will be randomized to receive either a deprescribing focused medication review or usual care.

The deprescribing focused medication therapy assessments will be done on half of the 143 residents residing on the second and third floors of the facility. The other half of residents will serve as the control group and continue to receive their annual medication review and regular care from the attending physicians and nurses.

The deprescribing intervention will be delivered by final year pharmacy students completing their practice experiences, under the supervision of clinical pharmacists at the LTC facility and clinical pharmacists from Memorial University's Medication Therapy Services (MTS) Clinic. Currently the clinic has a well developed procedure for providing in depth medication therapy reviews for residents of the community, upon referral by their primary care physician. Students will adapt this model of medication review to have a stronger deprescribing focus and be applicable to elderly residents of a LTC facility. The intervention will consist of an in depth medication therapy review with a focus on identifying any medications that may no longer be required or are deemed to be inappropriate or potentially unsafe in the elderly based on currently guidelines/criteria. The students will work closely with members of the resident's care team on a daily basis, as well as the resident and their family, to develop and implement a deprescribing plan.

ELIGIBILITY:
Inclusion Criteria (all of the following):

1. Over 65 years of age
2. Reside in St. Patrick's Mercy Home (2nd or 3rd floor units)

Exclusion Criteria (any of the following):

1. Do not take any regularly scheduled medications
2. Are receiving palliative care
3. Resident's physician or nursing team do not support participation
4. Resident or their substitute decision maker decline participation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Change in number of medications taken daily by residents | 3 and 6 months after receiving intervention
  Measured using facility medication logs and patient health records

SECONDARY OUTCOMES:
All cause mortality rate | 3 and 6 months after receiving the intervention
  Measured using patient health records
Instance of falls in the last 30 days | 3 and 6 months after receiving the intervention
  Measured using facility fall report logs
Frequency of emergency room visits, unplanned hospital admission and/or unplanned GP visits | 3 and 6 months after receiving the intervention
  Measured using patient health records
Cognitive function score | 3 and 6 months after receiving the intervention
  Measured using Cognitive Performance Scale (CPS) obtained from Resident Assessment Instrument (RAI) MDS 2.0
Bowel function | baseline, 3 and 6 months after receiving the intervention
  Measured using bowel chart data for the 14 days prior to the assessment date
Independence in activities of daily living | 3 and 6 months after receiving the intervention
  Measured using the Activities of Daily Living Scale (ADL) obtained from RAI MDS 2.0
Changes in general health | 3 and 6 months after receiving the intervention
  Measured using the Changes in Health, End-Stage Disease and Signs and Symptoms (CHESS) Score obtained from RAI MDS 2.0
Social engagement | 3 and 6 months after receiving the intervention
  Measured using Index of Social Engagement (ISE) Score obtained from RAI MDS 2.0
Aggressive behaviour | 3 and 6 months after receiving the intervention
  Measured using the Aggressive Behaviour Scale (ABS) obtained from RAI MDS 2.0
Frequency of pain | 3 and 6 months after receiving the intervention
  Measured using the Pain Scale obtained from RAI MDS 2.0

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Kelly, PharmD, Principal Investigator — Memorial University of Newfoundland
Locations (1):
- St Patrick's Mercy Home, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No